CLINICAL TRIAL: NCT03689309
Title: High Flow Oxygen During Spontaneous Breathing Trial in Patients With High Weaning Risk Failure: Impact on the Weaning Course at D7 From the First Spontaneous Breathing Trial. A Pilot Randomized Controlled Trial
Brief Title: High Flow Oxygen During Spontaneous Breathing Trial in Patients With High Weaning Risk Failure: Impact on the Weaning Course at D7 From the First Spontaneous Breathing Trial.
Acronym: ObiWEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHRO-2018-06
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Mechanical Ventilation; Mechanical Ventilator Weaning; Endotracheal Extubation
Keywords: Spontaneous breathing Trial; High Flow Oxygen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Classic SBT (C-SBT) (No Intervention): The patient is disconnected from the ventilator and remains 30 minutes without support but oxygen delivered through a heat humidifier filter that is usually connected on tracheotomy.
- 2. High Flow Oxygen SBT (HFO-SBT) (Experimental): The patient is disconnected from the ventilator and remains 30 minutes without support but high flow oxygen delivered through a dedicated piece that is usually connected on tracheotomy.
  Interventions: Procedure: High Flow Oxygen SBT

INTERVENTIONS:
Procedure: High Flow Oxygen SBT — The patient is disconnected from the ventilator and remains 30 minutes without support but high flow oxygen delivered through a dedicated piece that is usually connected on tracheotomy.
  Arms: 2. High Flow Oxygen SBT (HFO-SBT)

SUMMARY:
In intensive care unit (ICU), mechanical ventilation (MV) is part of routine care.

Weaning phase is a daily preoccupation for the caregivers. Prolonged MV can lead to many complications. Failing the weaning phase expose the patient to the need for reintubation, that improves the mortality.

The caregiver faces a major problem, in one hand the need to wean properly and quickly and on the other the risk of reintubation.

In order to help the clinician making the good choice, the spontaneous breathing trial (SBT) is a key tool. The international literature provides the investigators many ways to perform the SBT. The most common is the T-piece; the patient is disconnected from the ventilator and connected to a T-piece that can provide supplemental oxygen. Another one is the Support pressure trial, the patient is still connected to the ventilator, but the setups are changed to recreate the T-piece conditions.

In many French ICU's, the SBT is performed by using a heat humidifier filter that is directly connected to the endotracheal tube, this filter allows the clinician to provide supplemental oxygen in accordance with the patient need.

In high risk for reintubation patients, the SBT can create physical stress, that lead to prolonged MV.

In our ICU, for those patients, the investigators perform the SBT by connecting the patient to a device that provides high flow oxygen trough endotracheal connector for tracheotomy.

The investigators hypothesis that high flow oxygen SBT, will allow the high risk for reintubation patients to succeed the SBT.

DETAILED DESCRIPTION:
The investigators proposed to compare 2 strategies for SBT in high risk for reintubation patients:

1. Classic SBT (C-SBT)
2. High Flow Oxygen SBT (HFO-SBT)

This prospective randomized study had 2 conjoint primary outcome:

1. The HFO-SBT shows a better actuarial rate for extubation at day 7 from the begin of the weaning phase
2. Compare the reintubation rate at D7 from the extubation

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs.
* Admission in ICU
* Mechanically ventilated > 24 hours
* Mechanically ventilated using support ventilation mode
* Patient with one of these criterion:

  * Cardiac disease (left ventricular dysfunction LVEF <46%, antecedent of ischemic heart disease, antecedent of acute pulmonary edema)
  * Respiratory disease (COPD, Emphysema, bronchectiasis, asthma, obesity-hypoventilation syndrome, restrictive pulmonary disease)
* Informed and signed consent from the patient or next of kin.

Exclusion Criteria:

* Head trauma as a cause for ICU admission
* Neuromuscular disease prior ICU admission
* Tracheotomized patient
* Pregnancy
* Decision not to forgo life sustaining therapy
* Patient not affiliated with a social security organism
* Adult private from his liberty with judicial decision
* Patient that have already been included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Actuarial rate of extubation | Day 7
  This prospective randomized study had 2 conjoint primary outcomes to ensure the safety for the patients:
  1. The HFO-SBT shows a better actuarial rate for extubation at day 7 from the begin of the weaning phase
  2. Compare the reintubation rate at D7 from the extubation
  This prospective randomized study had 2 conjoint primary outcomes to ensure the safety for the patients:
  1. The HFO-SBT shows a better actuarial rate for extubation at day 7 from the begin of the weaning phase
  2. Compare the reintubation rate at D7 from the extubation
Reintubation Rate | Day 7
  This prospective randomized study had 2 conjoint primary outcomes to ensure the safety for the patients:
  1. The HFO-SBT shows a better actuarial rate for extubation at day 7 from the begin of the weaning phase
  2. Compare the reintubation rate at D7 from the extubation

SECONDARY OUTCOMES:
Success rate of the first SBT | Day 0
  Success rate of the first SBT will be compared between the two groups.
Ventilator free-days | Day 28
  Ventilator free-days at day 28 from the admission in ICU
Rate of Ventilator Associated Pneumonia | Day 7
  Rate of Ventilator Associated Pneumonia at day 7 from the extubation

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh NAY, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR d'Orleans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thille AW, Richard JC, Brochard L. The decision to extubate in the intensive care unit. Am J Respir Crit Care Med. 2013 Jun 15;187(12):1294-302. doi: 10.1164/rccm.201208-1523CI. PMID 23641924
- [Background] Ladeira MT, Vital FM, Andriolo RB, Andriolo BN, Atallah AN, Peccin MS. Pressure support versus T-tube for weaning from mechanical ventilation in adults. Cochrane Database Syst Rev. 2014 May 27;2014(5):CD006056. doi: 10.1002/14651858.CD006056.pub2. PMID 24865303
- [Background] Brochard L, Rauss A, Benito S, Conti G, Mancebo J, Rekik N, Gasparetto A, Lemaire F. Comparison of three methods of gradual withdrawal from ventilatory support during weaning from mechanical ventilation. Am J Respir Crit Care Med. 1994 Oct;150(4):896-903. doi: 10.1164/ajrccm.150.4.7921460.